CLINICAL TRIAL: NCT06770101
Title: Suicide Assessment and Feasible Evidence-based Treatments for Youth Living With HIV in Lilongwe: SAFETY Planning Pilot Trial
Brief Title: Suicide Assessment and Feasible Evidence-based Treatments for Youth Living With HIV in Lilongwe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Melissa Stockton, Assistant Professor of Psychiatry, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 857370; R34MH136204 (NIH)
Record Dates: First submitted 2025-01-09; First posted 2025-01-13 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: HIV; Suicide
Keywords: HIV; Suicide; Suicidal Ideation
MeSH Terms: conditions — Suicide; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: 2-arm individually randomized pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced Friendship Bench + Safety Planning (FB+SP) (Experimental): Friendship Bench (FB) problem-solving therapy and Safety Planning (SP)
  Interventions: Behavioral: Behavioral: Enhanced Friendship Bench + Safety Planning
- Augmented Usual Care (Active Comparator): Continue with usual outpatient care, augmented to provide mental health evaluation, brief supportive counseling, information, education and support on SIBs, and (if indicated) facilitation of referral to the clinic's psychiatric nurse or to Bwaila Hospital.
  Interventions: Behavioral: Augmented usual care

INTERVENTIONS:
Behavioral: Behavioral: Enhanced Friendship Bench + Safety Planning — The protocol will include six sessions, starting with the development of the SP during the first session. Each of the following sessions will include SIBs and suicide risk assessments, SP check-ins and revisions, as well as FB problem-solving to address SIBs and suicide risk. SP+FB will be delivered by selection of young counselors (mixed genders, aged 20-35) who are motivated to work with young people. Counseling sessions will take place in a discrete location within the HIV clinic and be available on weekends. Each structured session lasts 30-45 minutes and conducted in the participant's local language (Chichewa). After 4 sessions of individual therapy, the counselor can refer participants not improving or with suicidal ideation to a supervisor trained in mental health to reassess and manage the case. Case management may include additional counseling or pharmacotherapy, at the discretion of the managing clinician. Participants may also receive text message support and peer-support.
  Arms: Enhanced Friendship Bench + Safety Planning (FB+SP)
Behavioral: Augmented usual care — Care for suicidality in public facilities in Malawi includes options for basic supportive counseling by the primary provider or nurse, medication management by the primary provider, referral to the clinic's psychiatric nurse, or, for acute cases or crises, referral to the psychiatric units at tertiary care hospitals (Bwaila Hospital in Lilongwe District). Nurses and clinicians at the study sites have been specifically trained to use the Tool for Assessment of Suicide Risk for Adolescents (TASR-A) to assess ALWH considered at elevated risk for suicide. For this study, usual care will be augmented by a trained study nurse who will provide mental health evaluation, brief supportive counseling, information, education and support on SIBs, and (if indicated) facilitation of referral to the clinic's psychiatric nurse or to Bwaila Hospital.
  Arms: Augmented Usual Care

SUMMARY:
The overall aim of this study is to determine the feasibility, fidelity, acceptability, and preliminary effectiveness of the Friendship Bench +Safety Planning intervention in reducing suicidal ideation and behaviors (SIBs) and improving HIV engagement amongst adolescents living with HIV (ALWH) when compared to augmented usual care.

DETAILED DESCRIPTION:
This project aims to evaluate the feasibility, acceptability, fidelity, and preliminary effectiveness of the enhanced Friendship Bench+Safety Planning (FB+SP) intervention model. We will enroll 60 depressed ALWH who report suicidality from four facilities in Lilongwe, Malawi, and randomize them 1:1 to the enhanced FB+SP model or augmented usual care. This pilot trial is a step toward our long-term goal of generating and implementing an evidence-based model to prevent suicide in Malawi amongst ALWH by enhancing the capacity of the health system to identify suicidality and provide evidence-based care. Information gathered in this proposal will be used to develop a subsequent randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-19
* Diagnosed with HIV
* Report current or historical suicidal ideation and behaviors (SIBs) on question 9 of the Patient Health Questionnaire modified for adolescents (PHQ-9-A) and the Ask Suicide-Screening questionnaire (ASQ)
* Living in the clinic's catchment area with intention to remain for more than 1 year
* Willing to provide consent (age 18+ or 16-17 years old and married and thereby considered emancipated minors per Malawi law) or assent with parental consent (age 13-17).

Exclusion Criteria:

* Refuse to participate
* Refuse to be audio-taped for in-depth interviews

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-14 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Study retention (study feasibility) | Through study completion- 6 months
  This outcome measure of feasibility will be measured as the ability to retain ALWH in the pilot trial. Feasibility will be evaluated by measuring the number of participants retained in the study (number of patients enrolled at baseline who are still enrolled in the trial) through study completion.
Recruitment rate (Intervention feasibility) | Baseline
  This outcome measure of feasibility will be measured as the ability to successfully enroll ALWH in the pilot trial. Feasibility will be evaluated by measuring the recruitment rate (number of patients approached in order to accrue the final sample).
Overall satisfaction with the intervention among participants (intervention acceptability) | 6 months
  The proportion of participants who found the intervention acceptable and helpful among all participants who received the intervention.
Proportion of sessions meeting fidelity threshold (intervention fidelity) | 6 months
  The proportion of sessions meeting or exceeding expectations for at least 80% of the total number of fidelity checklist items assessed per session during random monitoring sessions out of all sessions monitored.

SECONDARY OUTCOMES:
Prevalence of suicidal ideation and behaviors | 6 months
  The proportion of participants in each arm who report experiencing suicidal ideation and behaviors out of all participants in that arm. Suicidal ideation and behaviors will be documented using question 9 of the Patient Health Questionnaire-9 modified for Adolescents (PHQ-A), which is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression with scores ranging from 0 to 27, where higher scores indicate greater self-reported depression and the Ask Suicide-Screening Questions (ASQ), which is a brief screening tool of five yes/no items addressing suicide risk.
Prevalence of suicide risk | 6 months
  The proportion of participants in each arm with passive to active suicide risk out of all participants in that arm. Suicide risk will be measured using the study's Suicide Risk Assessment Protocol.
Prevalence of depressive symptoms | 6 months
  The proportion of participants in each arm who report elevated depressive symptoms out of all participants in that arm. Depressive symptoms will be measured using the Patient Health Questionnaire-9 modified for Adolescents (PHQ-A) which is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression with scores ranging from 0 to 27, where higher scores indicate greater self-reported depression.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Stockton, PhD, Principal Investigator — University of Pennsylvania
Locations (4):
- Malawi (4):
  - Area 18 Health Center, Lilongwe
  - Area 25 Health Center, Lilongwe
  - Kawale Health Center, Lilongwe
  - Lighthouse Health Center, Lilongwe

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be posted to the National Insititute of Mental Health (NIMH) Data Archive pursuant to the requirements of that site.

REFERENCES:
- [Derived] Stockton MA, Waddell K, Mphonda SM, Bhushan NL, January J, Masulani C, Brown G, Udedi MM, Pence BW, Chiwanda J, Gaynes BN, Kulisewa K. Suicide assessment and feasible evidence-based treatments for adolescents living with HIV in Malawi: Protocol for a pilot randomized controlled trial. PLoS One. 2025 Sep 3;20(9):e0330847. doi: 10.1371/journal.pone.0330847. eCollection 2025. PMID 40901775